CLINICAL TRIAL: NCT03580798
Title: Ridge Preservation Comparing the Traditional Approach vs. Early Implant Placement With Simultaneous Contour Augmentation
Brief Title: Ridge Preservation Comparing Simultaneous vs. Delayed Grafting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients available
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Director of Graduate Peridontics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18.0348
Record Dates: First submitted 2018-06-13; First posted 2018-07-09 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Grafting (Experimental): 8 weeks after extraction implant placement and simultaneous osseous grafting.
  Interventions: Procedure: Delayed graft
- Simultaneous Grafting (Active Comparator): At the time of extraction the socket will be grafted and implant placed 4 months later.
  Interventions: Procedure: Simultaneous graft

INTERVENTIONS:
Procedure: Delayed graft — 8 weeks post-extraction 15 test patients will receive implant placement plus osseous grafting.
  Arms: Delayed Grafting
Procedure: Simultaneous graft — At the time of extraction osseous graft will be placed in the socket and implant placed 4 months later.
  Arms: Simultaneous Grafting

SUMMARY:
Comparison of the clinical healing of simultaneous vs. delayed grafting for dental implant placement.

DETAILED DESCRIPTION:
The primary aims of this study are to compare the clinical and histologic results of a traditional ridge preservation with implant placement at 16 weeks (control group) with early implant placement (8 weeks) with simultaneous contour augmentation as described by Buser (test group).

ELIGIBILITY:
Inclusion Criteria:

* Have one non-molar maxillary tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by 2 teeth.
* Healthy persons at least 18 years old.
* Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

* Patients with debilitating systemic disease, or diseases that have a clinically significant effect on the periodontium.
* Exclude any molar tooth.
* Presence of or history of osteonecrosis of jaws.
* Patients with current or previous history of IV bisphosphonates, irrespective of duration.
* Patients taking oral bisphosphonates for ≥ 3 years.
* Pregnant women.
* Allergy to any material or medication used in the study.
* Patients who need prophylactic antibiotics prior to dental procedures.
* Previous head and neck radiation therapy.
* Chemotherapy in the previous 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Final ridge width for simultaneous and delayed grafting treatment. | 16 to 20 weeks
  Measure final ridge width to determine if adequate bone is available.

SECONDARY OUTCOMES:
Soft tissue thickness | 16 to 20 weeks
  Facial and occlusal
Histology | 16 weeks
  Histologic composition for control group only
Implant dehiscence | 20 weeks
  Implant dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics, UofL School of Dentistry, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No